CLINICAL TRIAL: NCT02815332
Title: A Randomized, Double-blind, Vehicle Controlled Study to Assess the Safety and Efficacy of BPX-01 Minocycline Topical Gel in the Treatment of Moderate to Severe Inflammatory Acne Vulgaris
Brief Title: BPX-01 Minocycline Topical Gel in the Treatment of Acne Vulgaris
Acronym: OPAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPX-01-C03
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BPX-01 Vehicle Topical Gel (Placebo Comparator): Approximately 1 gram applied once daily for 12 weeks
  Interventions: Drug: BPX-01 Vehicle Topical Gel
- BPX-01 1% Minocycline Topical Gel (Experimental): Approximately 1 gram applied once daily for 12 weeks
  Interventions: Drug: BPX-01 1% Minocycline Topical Gel
- BPX-01 2% Minocycline Topical Gel (Experimental): Approximately 1 gram applied once daily for 12 weeks
  Interventions: Drug: BPX-01 2% Minocycline Topical Gel

INTERVENTIONS:
Drug: BPX-01 1% Minocycline Topical Gel — Approximately 1 gram applied once daily for 12 weeks
  Other Names: BPX-01 Topical Gel
  Arms: BPX-01 1% Minocycline Topical Gel
Drug: BPX-01 2% Minocycline Topical Gel — Approximately 1 gram applied once daily for 12 weeks
  Other Names: BPX-01 Topical Gel
  Arms: BPX-01 2% Minocycline Topical Gel
Drug: BPX-01 Vehicle Topical Gel — Approximately 1 gram applied once daily for 12 weeks
  Other Names: BPX-01 Vehicle Gel
  Arms: BPX-01 Vehicle Topical Gel

SUMMARY:
This is a 12-week, multi-center, double-blind, randomized, three-arm, vehicle-controlled study.

Subjects will be randomized (1:1:1) to 1% or 2 % BPX-01 gel, or vehicle. Subjects will apply 1g of the gel as a thin film to the entire face at least 30 minutes before bedtime each night for 12 weeks. Lesion counts, IGA, and Patient-Reported Outcomes (PGI-S and PGI-I) will be performed to assess efficacy.

Blood draws will be collected at baseline (Day 0), and at Weeks 4 and 12 to evaluate the level of minocycline in plasma. Safety will be assessed with the vital signs, brief physical examination, clinical laboratory tests, cutaneous tolerance score, incidence of minocycline-induced skin hyperpigmentation, incidence of visual disturbances and/or headaches suggestive of pseudotumor cerebri, and collection of adverse events.

DETAILED DESCRIPTION:
This is a phase 2b, randomized, double-blind, vehicle-controlled study to Assess the Safety and Efficacy of BPX-01 Minocycline Topical Gel in the Treatment of Moderate to Severe Inflammatory Acne Vulgaris.

Study Population: Approximately 225 male or female subjects aged between 9 and 40 years with moderate to severe inflammatory non-nodular acne vulgaris will be included in this study.

Number of Sites: Approximately 15 centers from the United States will participate in this study.

Study Duration: Overall study duration is expected to be approximately 24 weeks (6 months). The study duration for individual subjects is approximately 16 weeks (including the screening period).

Hypothesis: BPX-01 improves disease condition in subjects with moderate to severe inflammatory non-nodular acne vulgaris compared with vehicle.

Objectives:

Primary:

* To evaluate the efficacy of BPX-01 minocycline 1% or 2% topical gel in the treatment of inflammatory non-nodular acne vulgaris

Secondary:

* To evaluate the plasma level of minocycline after once daily application of 1% or 2% BPX 01 topical gel
* To evaluate the safety of BPX-01 minocycline 1% or 2% topical gel

Endpoints:

Primary Efficacy Endpoint:

* Absolute mean change from baseline in inflammatory lesion counts at Week 12

Secondary Efficacy Endpoint:

* Proportion of subjects with at least a two-grade reduction in IGA at Week 12

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 9 and 40 years of age.
2. Subjects do not have any medical conditions, other than acne vulgaris, that in the opinion of the investigator, put the subject at unacceptable risk or could interfere with study assessments or integrity of the data.
3. Moderate to severe inflammatory non-nodular acne vulgaris.
4. Female subjects of childbearing potential (including pre-puberty) are willing to use effective contraceptive method for at least 28 days before baseline (Day 0) and at least 28 days after the last study product administration or have a sterilized or same-sex partner for the duration of the study.
5. Treatment with hormonal therapy must be on a stable dose and frequency for at least 12 weeks before baseline (Day 0) and must remain stable throughout the study.
6. Subjects who use make-up, facial moisturizers, creams, or lotions, cleansers and/or sunscreens must have used the same product brands/types for a minimum period of 14 days prior to baseline (Day 0), must agree not to change brand/type or frequency of use throughout the study and must agree not to use make-up, facial moisturizers, creams, or lotions, cleansers and/or sunscreens on the clinic visit days before the visit.
7. Subjects must be capable of giving informed consent and the written informed consent must be obtained prior to any study-related procedures. Subject under 18 years of age must sign an assent form, and their parent(s) or legal representative must have read and signed the informed consent form prior to any study-related procedures.

Exclusion Criteria:

1. Female subject who is breastfeeding, pregnant or who is planning a pregnancy during the study.
2. Have acne fulminans or conglobata, or nodulocystic acne.
3. Have a history of skin disease, presence of skin condition, or excessive facial hair that, in the opinion of the investigator, would interfere with the study.
4. Have a history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
5. Have a history of minocycline-induced hepatitis, minocycline-induced arthritis, minocycline-induced lupus or minocycline/tetracycline-induced pseudotumor cerebri.
6. Presence of minocycline-induced hyperpigmentation at screening or baseline (Day 0).
7. Presence of visual disturbances and/or headaches suggestive of pseudotumor cerebri at screening or baseline (Day 0).
8. Have a clinical chemistry or hematology laboratory value that is abnormal at the screening visit and that is considered clinically significant by the investigator.
9. Has an ALT or AST at screening greater than or equal to 2 times the upper limit of normal.
10. Have used on the face an over-the-counter (OTC) topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, salicylic acid, α-hydroxy/glycolic, antibacterial/antiseptic soap or wash within 14 days prior to baseline (Day 0).
11. Have used prescription topical retinoid (e.g. tretinoin, tazarotene, adapalene) or antimicrobials (e.g. clindamycin, erythromycin) or other prescription topical medications for the treatment of acne vulgaris within 28 days of baseline (Day 0).
12. Have used systemic antibiotics or other systemic anti-acne drugs not mentioned in the exclusion criteria within 28 days of baseline (Day 0).
13. Have used oral, intranasal, or injectable corticosteroids within 28 days of baseline (Day 0) or require them during the study. Inhaled corticosteroids for stable medical conditions are allowed.
14. Have received an investigational therapy (including investigational drug or procedure) within 28 days of baseline (Day 0) or plan to use one during the study.
15. Have had a facial procedure (e.g. chemical peel, laser, microdermabrasion) within 8 weeks of baseline (Day 0).
16. Have excessive sun exposure, is planning a trip to a sunny climate or used tanning booths within 28 days prior to baseline (Day 0) or is not willing to minimize natural and artificial sunlight exposure during the study.
17. Have received photodynamic therapy or phototherapy with blue or red light within 12 weeks of baseline (Day 0).
18. Have used androgen receptor blockers (such as spironolactone or flutamide) within 12 weeks of baseline (Day 0).
19. Have used drospirenone, chlormadinone acetate, and cyproterone acetate within 26 weeks of baseline (Day 0).
20. Have used oral retinoid (e.g., isotretinoin) within 52 weeks prior to baseline (Day 0) or vitamin A supplements greater than 10,000 U/d within 26 weeks of baseline (Day 0).
21. History of clinically significant drug or alcohol abuse in the last year prior to baseline (Day 0) as judged by the investigator.
22. Has known or suspected allergy to minocycline, tetracycline-class antibiotics or any component of the investigational product.

Ages: 9 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | 12 weeks
  Absolute mean change from baseline in inflammatory lesion counts

SECONDARY OUTCOMES:
Reduction in IGA | 12 weeks
  Proportion of subjects with at least a two-grade reduction in IGA from baseline

CONTACTS AND LOCATIONS:
Overall Officials: AnnaMarie Daniels, Study Director — Sponsor (BioPharmX)
Locations (15):
- United States (15):
  - Santa Monica, California
  - Coral Gables, Florida
  - Lake Mary, Florida
  - Newnan, Georgia
  - Louisville, Kentucky
  - Las Vegas, Nevada
  - Montclair, New Jersey
  - New York, New York
  - Highpoint, North Carolina
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Pflugerville, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes